CLINICAL TRIAL: NCT02536950
Title: An Outpatient Study of Automated Blood Glucose Control With an Insulin-Only Bionic Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce A. Buckingham (Other)
Collaborators: Boston University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Bruce A. Buckingham, Professor of Pediatrics (Endocrinology), MD, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Device Feasibility
Other Study IDs: IRB34914
Record Dates: First submitted 2015-07-18; First posted 2015-09-01 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: bionic pancreas; closed-loop control; artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Blinded Sensor (No Intervention): Subjects will wear a blinded Dexcom G4P (Generation 4 Platinum) AP (Artificial Pancreas) glucose sensor for a week
- Fixed set point (Experimental): Subjects will be in a hotel and use a fixed set point for glucose control for two days initialized at 130 mg/dl. The setpoint will be adjusted, if necessary, over the two days in the hotel before they are sent home for 5 days
  Interventions: Device: Fixed set point
- Variable Set Point (Experimental): Subjects will begin using a "variable" setpoint which will make adjustments based on their past glucose control over the previous day
  Interventions: Device: Variable set point

INTERVENTIONS:
Device: Fixed set point — Fixed set point arm: A fixed setpoint will be used initially. Staff will observe glucose control over 2 days while subjects remain in a hotel environment, and then over 5 more days in the same subjects in an outpatient setting. The clinical staff will adjust this target up or down by 15 mg/dl based on their glycemic control in the hotel setting.
  Arms: Fixed set point
Device: Variable set point — Variable set point arm: The setpoint will be variable over a 30 mg/dl range and glycemic control will be optimized based on the preceding 24-hour window.
  Arms: Variable Set Point

SUMMARY:
This is an open-label, non-randomized, pilot study to determine the safety and feasibility of the insulin-only bionic pancreas.

DETAILED DESCRIPTION:
A total of 16 subjects, ages 18-45, will be enrolled in this crossover study. The study will consist of three 7-day study arms in the following order, one usual care arm, one bionic pancreas insulin only arm with a static glucose target, and one bionic pancreas insulin only arm with at dynamic glucose target.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 1 year
* insulin pump for ≥ 6 months
* Prescription medication regimen stable for > 1 month
* Subject comprehends written English
* Female patients who are sexually active must be on acceptable method of contraception e.g. oral contraceptive pill, diaphragm, IUD (Intrauterine Device)
* Female patients must have a negative urine pregnancy test
* Informed Consent Form signed by the subject
* Lives and works within a 60 minute drive-time radius of Stanford University
* Willing to remain within a 60 minute drive-time radius of Stanford University during all 3 of the 7-day study arms (21 days)
* Have someone over 18 years of age who lives with them,

Exclusion Criteria:

* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days), use of marijuana within 1 month of enrollment, or other substance abuse (use within the last 6 months of controlled substances other than marijuana without a prescription)
* Subject has a history of diagnosed medical eating disorder
* Subject has a history of visual impairment which would not allow subject to participate
* Subject has an active skin condition that would affect sensor placement
* Subject has adhesive allergies
* Subjects requiring an intermediate or long-acting insulin (such as NPH, Neutral Protamine Hagedorn, detemir or glargine)
* Subjects requiring other anti-diabetic medications other than insulin (oral or injectable)
* Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
* Unwilling or unable to refrain from drinking more than 2 drinks in an hour or more than 4 drinks in a day or use of marijuana during the trial
* Subject has active Graves' disease
* Subjects with inadequately treated thyroid disease or celiac disease
* History of liver disease Renal failure on dialysis
* Personal history of cystic fibrosis, pancreatitis, pancreatic tumor, or any other pancreatic disease besides type 1 diabetes
* Any known history of coronary artery disease
* Abnormal EKG (electrocardiogram) consistent with coronary artery disease or increased risk of malignant arrhythmia
* Congestive heart failure (established history of congestive heart failure , lower extremity edema, paroxysmal nocturnal dyspnea, or orthopnea)
* History of transient ischemic attack (TIA) or stroke
* Seizure disorder, history of any non-hypoglycemic seizure within the last two years, or ongoing treatment with anticonvulsants
* History of hypoglycemic seizures (grand-mal) or coma in the last year
* History of pheochromocytoma:
* episodic or treatment refractory (requiring 4 or more medications to achieve normotension) hypertension
* paroxysms of tachycardia, pallor, or headache
* personal or family history of MEN 2A (multiple endocrine neoplasia), MEN 2B, neurofibromatosis, or von Hippel-Lindau disease
* History of adrenal disease or tumor
* Hypertension with systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 despite treatment
* Untreated or inadequately treated mental illness
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
* Unable to completely avoid acetaminophen for duration of study
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study
* History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
* History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
* Lives in or frequents areas with poor Verizon wireless network coverage (which would prevent remote monitoring)
* Any factors that, in the opinion of the site principal investigator or overall principal investigator, would interfere with the safe completion of the study

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mean glucose | change over 5 days
  Dexcom G4P AP mean glucose

SECONDARY OUTCOMES:
% time <50 mg/dl | change over 5 days
  Fraction of Dexcom G4P AP readings <60 mg/dl
% time <70 mg/dl | change over 5 days
  Fraction of Dexcom G4P AP readings <70 mg/dl
% time 70-120 mg/dl | change over 5 days
  Fraction of Dexcom G4P AP readings 70-120 mg/dl
% time 70-180 mg/dl | change over 5 days
  Fraction of Dexcom G4P AP readings 70-180 mg/dl
% time >180 mg/dl | change over 5 days
  Fraction of Dexcom G4P AP readings >180 mg/dl
% time >250 mg/dl | change over 5 days
  Fraction of Dexcom G4P AP readings >250 mg/dl
% time < 60 mg/dl | Change over 5 days
  Fraction of Dexcom G4AP readings < 60 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Buckingham, MD, Principal Investigator — Stanford School of Medicine, Pediatric Endocrinology
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No